CLINICAL TRIAL: NCT00328094
Title: Impact of Tight Control of Perioperative Blood Glucose in Patients Undergoing Vascular Surgery on Their Perioperative Cardiovascular and Overall Morbidity and Mortality
Brief Title: Glycemic Control to Prevent Cardiac Morbidity in Vascular Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The recruitment rate slowed considerably
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Balachundhar Subramaniam, Staff Anesthesiologist, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2005P-000299
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Results first posted 2013-04-09 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Peripheral Vascular Disease; Abdominal Aortic Aneurysm
Keywords: Tight; Glycemic; control; outcomes; peripheral vascular disease; infection; cardiovascular; morbidity; mortality
MeSH Terms: conditions — Peripheral Vascular Diseases; Aortic Aneurysm, Abdominal; Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CII, Continuous Insulin Infusion (Experimental): Continuous intravenous insulin infusion to control glucose to <150 mg/dL in patients undergoing open peripheral vascular bypass surgery
  Interventions: Drug: continuous intravenous insulin infusion
- IIB, Intermittent insulin boluses (Active Comparator): Intermittent intravenous insulin insulin boluses to a blood glucose target of <150mg/dL in patients undergoing peripheral vascular bypass surgery
  Interventions: Drug: continuous intravenous insulin infusion

INTERVENTIONS:
Drug: continuous intravenous insulin infusion — Tight glucose control versus standard of care
  Other Names: CII-continuous insulin infusion; II-Intermittent insulin boluses

SUMMARY:
Aggressive intraoperative and postoperative management of blood glucose may substantially decrease perioperative cardiovascular and infectious complications in diabetic and non-diabetic patients undergoing vascular surgery.

The purpose of this study is to compare the tight versus traditional blood glucose control in diabetics and non-diabetics undergoing vascular surgery in regard to their postoperative fatal and nonfatal cardiac outcomes, and the secondary effects such as rate of infections, overall morbidity and 30-day mortality.

DETAILED DESCRIPTION:
This is a randomized, prospective controlled trial in both diabetic and non diabetic patients undergoing vascular surgery such as abdominal aortic, infra inguinal vascular bypass procedures and amputations, comparing tight versus standard blood glucose control regimens in the operating room, post anesthesia care unit and in the postoperative vascular intensive care unit up to 48 hours and its impact on the cardiovascular, infectious and other morbidity and mortality during the hospital admission and up to 30 days from surgery.

After obtaining informed consent, the study subjects will be randomized to tight versus standard blood glucose control regimens. These regimens will be started in the operating room and continued for the first 48 hours or until their discharge, whichever is earlier. All the patients will be inpatients. Day surgery patients will be excluded.

The anesthesiologist providing patient care will be given either the tight glucose control protocol or the standard sliding scale insulin protocol. In the tight control regimen, target blood glucose is 100-150 mg/dl. If 3 consecutive blood glucose (BG) level >150 mg/dL or 1 BG level >200 mg/dL, then the insulin infusion will be initiated in the tight control group. The insulin infusion rate adjustments will be made based on the blood sugar results. In post anesthetic care unit (PACU) and vascular intensive care unit (VICU), these protocols will be nurse driven. The adjustments will be made based on the current blood sugar levels as well as the insulin infusion rates. They are adjusted in such a way to account for the rate of change of blood sugars and the presence of steroid therapy in the patients. The frequency of blood glucose testing in this group will be every 1-hour until stable (when frequent changes in insulin dosage are no longer necessary, and glucose is in the range of 100 to 150 for 3 consecutive blood sugar checks); then test every 2 hours for 3 consecutive target values and then every 4 hours thereafter. If there is a change in the infusion rates, then blood sugar checks will be done every hour and the cycle followed thereafter.

In the standard sliding scale insulin group, blood sugars will be treated with insulin boluses if the blood sugars go more than 150 mg/dL and blood glucose will be monitored every 4 hours.

These regimens will be initiated after 2 weeks of in-service training for anesthesiologists, post anesthetic care unit (PACU) and vascular intensive care unit (VICU) nurses. The study investigators will provide this training. Insulin infusion in the tight control regimen will be started through pump piggyback to maintenance intravenous infusion as follows. Insulin infusion bags will be made by the pharmacy (100 units in a 100 ml bag). The anesthesiologists in the operating room and PACU, and VICU nurses will perform blood glucose monitoring, bolus insulin administration, and infusion initiation and rate adjustments as specified by the protocol. Blood glucose levels will be tested by finger stick method or arterial line drop sample.

ELIGIBILITY:
Inclusion Criteria:

* Abdominal aortic surgery
* Supra and infrainguinal peripheral vascular bypass surgery
* Below knee amputations
* Above knee amputations
* Diabetics and nondiabetics
* American Society of Anesthesiologists (ASA) I-III

Exclusion Criteria:

* Brittle diabetics
* ASA 1V,V
* Second surgery in same admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2006-03; Primary Completion 2008-04 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Balachundhar Subramaniam, Principal Investigator — Beth Israel Deaconess Medical Center, Boston MA
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Furnary AP, Zerr KJ, Grunkemeier GL, Starr A. Continuous intravenous insulin infusion reduces the incidence of deep sternal wound infection in diabetic patients after cardiac surgical procedures. Ann Thorac Surg. 1999 Feb;67(2):352-60; discussion 360-2. doi: 10.1016/s0003-4975(99)00014-4. PMID 10197653
- [Background] van den Berghe G, Wouters P, Weekers F, Verwaest C, Bruyninckx F, Schetz M, Vlasselaers D, Ferdinande P, Lauwers P, Bouillon R. Intensive insulin therapy in critically ill patients. N Engl J Med. 2001 Nov 8;345(19):1359-67. doi: 10.1056/NEJMoa011300. PMID 11794168
- [Background] Zimmerman CR, Mlynarek ME, Jordan JA, Rajda CA, Horst HM. An insulin infusion protocol in critically ill cardiothoracic surgery patients. Ann Pharmacother. 2004 Jul-Aug;38(7-8):1123-9. doi: 10.1345/aph.1E018. Epub 2004 May 18. PMID 15150382
- [Background] Kersten JR, Warltier DC, Pagel PS. Aggressive control of intraoperative blood glucose concentration: a shifting paradigm? Anesthesiology. 2005 Oct;103(4):677-8. doi: 10.1097/00000542-200510000-00002. No abstract available. PMID 16192757

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Perioperative period in Beth Israel Deaconess Medical Center, West Campus was the only location for the recruitment.
Pre-assignment Details: 252 were assessed for eligibility. 10 did not meet inclusion criterion.
Groups:
- Continuous Insulin Infusion: Tight glucose group with insulin infusion
- Intermittent Insulin Bolus: Intermittent insulin boluses group
Period: Overall Study
Arm/Group | Continuous Insulin Infusion | Intermittent Insulin Bolus
Started | 117 | 125
Completed | 114 (2 did not receive intervention. 1 patient refusal) | 122 (3 did not receive interevention. 1 post induction arrest. 1 case cancelled.)
Not Completed | 3 | 3
Not completed — Physician Decision | 3 | 3

BASELINE CHARACTERISTICS:
Population: assessed for eligibility 252. 10 were found ineligible. 242 were randomized.6 patients did not receive interventions they were supposed to. Total number of patients analyzed were 236.
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Insulin Infusion | Intermittent Insulin Bolus | Total
Number analyzed (Participants) | 114 | 122 | 236
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 43 | 92
  >=65 years | 65 | 79 | 144
Age Continuous [Mean (Standard Deviation); unit: years] | 67 (10) | 71 (11) | 69 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 56 | 103
  Male | 67 | 66 | 133
Region of Enrollment [Number; unit: participants]
  United States | 114 | 122 | 236

OUTCOME MEASURES:

1. Secondary Outcome: Incidence of Wound Infections
Time Frame: postoperative
Measure: Number; unit: participants
Arm/Group | Continuous Insulin Infusion | Intermittent Insulin Bolus
Number analyzed (Participants) | 114 | 122
participants | 35 | 29
Statistical Analysis 1: Comparison: Continuous Insulin Infusion vs Intermittent Insulin Bolus; Test type: Superiority or Other; p = 0.23, Chi-squared; Risk Ratio (RR) = 1.29, 95% CI 2-sided [0.85 to 1.97]

2. Primary Outcome: Composite (Myocardial Infarction and CHF)
Time Frame: hospital length of stay
Measure: Number; unit: Number of patients
Arm/Group | Continuous Insulin Infusion | Intermittent Insulin Bolus
Number analyzed (Participants) | 114 | 122
Number of patients | 4 | 15

ADVERSE EVENTS:
Time Frame: Study period. Hospital stay
Arm/Group | Continuous Insulin Infusion | Intermittent Insulin Bolus
Serious Adverse Events (participants affected / at risk) | 10/114 | 5/122
Other Adverse Events (participants affected / at risk) | 23/114 | 22/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous Insulin Infusion (N=114) | Intermittent Insulin Bolus (N=122)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 10 (10) | 5 (5) — Blood glucose < 60 mg/dL atleast once
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous Insulin Infusion (N=114) | Intermittent Insulin Bolus (N=122)
Creatinine > 25% increase (Renal and urinary disorders) | 23 (23) | 22 (22) — INcrease in creatinine > 25% in the postoperative period from the preoperative period

LIMITATIONS AND CAVEATS:
A trial to adequately address mortality would require 5000 to 6000 patients. The alpha levels for significance were not adjusted for the interim analyses because of the unplanned issues with subject recruitement as surgery became percutaneous.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes